CLINICAL TRIAL: NCT06139497
Title: Feasibility and Effectiveness of a Pilot Program of Physical Activity to Improve Functional Limitations and Disability in HIV-infected Adults Older Than 50 From Côte d'Ivoire
Brief Title: Implementation and Effectiveness of Physical Activity to Prevent Disability in HIV-infected Adults Older Than 50 From Côte d'Ivoire
Acronym: VIRAGE+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut de Recherche pour le Développement (IRD) (Unknown); Programme PAC-CI (Unknown); Université Paris Cité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANRS 0396 VIRAGE+
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Cardiovascular Diseases; Insulin Resistance Syndrome X
Keywords: HIV; Disabilities; Aging; Readaptation; Resource-limited countries; Physical activity; non-communicable disease
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases; Metabolic Syndrome; Motor Activity; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Hybrid type 2 (dual focus on effectiveness and implementation outcomes)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Groupes-based arm (Experimental): Participants are invited to participate in group sessions directly supervised by a coach. The other sessions are unsupervised. During the first 24 weeks (active phase), the supervised group sessions are scheduled on a weekly basis while they are more spaced out, on a monthly basis, during the second part of the 48 weeks (maintenance phase).
  Interventions: Behavioral: Physical activity programme
- Home-based arm (Experimental): Participants have to perform the same exercise programme at home. Start with two weeks of direct supervision to learn how to carry out safely the training and how to adapt the intensity of the exercise using the rated perceived exertion (RPE) and the heart rate self-monitored during exercise.
  Interventions: Behavioral: Home-based physical activity
- Control arm (No Intervention): Health education session every months.

INTERVENTIONS:
Behavioral: Physical activity programme — 48-week exercise programme including aerobic, resistance, balance and flexibility exercises twice to three times per week. The sessions are supervised by a coach at least once a week during the first 6 months then monthly. The other session of the PA programme is performed at home and the overall weekly PA is reviewed with the coach at the end of the supervised session.
  Arms: Groupes-based arm
Behavioral: Home-based physical activity — 48-week exercise programme including aerobic, resistance, balance and flexibility exercises twice to three times per week. Participants have to perform the exercise programme at home exclusively. They are called every week by a research assistant to review the activities performed, collect information on their adherence and perception on the programme.
  Arms: Home-based arm

SUMMARY:
The overall objective of this research is to provide evidence on the effectiveness and implementation of two strategies deliver a structured programme of physical activity (PA) people living with HIV older than 50 years from Ivory Coast.

The research will starts a baseline formative research including people with and without HIV infection.

Participants are randomized 1:1:1 to one for the following group: (1) a reference arm receiving a group-based PA program supervised by a coach (n = 60), (2) an exploratory arm receiving a home-based PA program with remote supervision via phone calls and messaging apps (n = 60) and (3) a control arm receiving health education sessions (n = 60). The total follow-up period is 12 months, with an initial 6-month active phase and then a 6-month maintenance.

The primary effectiveness outcome is the improvement at the 6-minute step-up test between baseline and 6 months. Secondary outcomes include changes in performance on other functional tests and improvement of cardio-metabolic risk factors. Implementation outcomes include acceptability, adoption, feasibility and sustainability of the intervention.Implementation outcomes will be assessed using mixed methods during the intervention. Effectiveness outcomes and patient-centered outcomes will be assessed at baseline, 6 and 12 months.

DETAILED DESCRIPTION:
This is is a prospective, randomised, pilot trial with two phases: a 6-month active phase to implement the intervention and a 6-month maintenance phase to evaluate the sustainability of the intervention's effects. This study adopts a type II hybrid design assessing both the effectiveness of the intervention and the implementation outcomes to identify factors influencing its adoption by users, as well as its integration into healthcare practices

It starts with a baseline research combining a cross-sectional study and a qualitative formative research. The cross-sectional study comprises clinical evaluations, functional tests, as well as quantitative evaluations by questionnaire of disability (WHODAS, HDQ) and depression (PHQ-9). It includes 300 people living wiht HIV (PLHIV) receiving antiretroviral therapy and followed at the Avocatier health facility (FSU) and the El Rapha medical health centre (CMS), in the Abobo district, Abidjan. A comparison group of adults without HIV infection of similar sex and age distribution is included as a reference group (n = 150).

The qualitative research explores how the practice of physical activity is perceived culturally and socially and to determine the factors that may influence the implementation of this type of activity.

The intervention consists of a 48-week exercise programme including aerobic, resistance, balance and flexibility exercises twice to three times a week for at least 60 minutes. Two delivery approaches for the exercise programme are proposed. In the group-based arm, participants are invited to participate in group sessions directly supervised by a coach. The other sessions are unsupervised. During the first 24 weeks (active phase), the supervised group sessions are scheduled on a weekly basis while they are more spaced out, on a monthly basis, during the second part of the 48 weeks (maintenance phase). In the home-based arm, participants have to perform the same exercise programme at home. Participants are contacted by phone by a study staff every week to review the activities performed, collect information on their adherence to and perception of the programme and to provide positive feedback, help to addess challenges and reinforce their motivation. Participants of the control group are offered monthly health education sessions and a delayed participation to the programme.

ELIGIBILITY:
Eligibility criteria for the intervention :

Inclusion criteria:

* Age ≥50 years
* Documented HIV infection.
* Receiving antiretroviral therapy for ≥ 12 months.
* Residing in the Abobo district (Côte d'Ivoire).
* Presence of at least one functional limitation or disability criterion among the following:

  * Performance in the 6-minute walk test ≤ 300 m.
  * Handgrip strength ≤ 35 kg for men or ≤ 24 kg for women.
  * WHODAS score ≥ 10.
  * SPPB score between 4 and 9.
* Signed informed consent.

Exclusion criteria

* Medical contraindication to physical activity.
* Anticipated unavailability.
* Severe functional limitation (SPPB ≤ 3).
* Another health condition requiring priority care.

Eligibility criteria for the formative research:

Inclusion criteria:

People living with HIV:

* Age ≥40 years
* Documented HIV infection.
* Receiving antiretroviral therapy for ≥ 12 months.

Controls:

* Age ≥40 years
* Negative HIV test within the last 12 months;
* Living in Abobo area
* Written consent to participate to the study

Exclusion Criteria:

Participants living with HIV:

* HIV infection with HIV-2 type only
* Any clinical symptoms suggesting an acute infection
* Any life-threatening pathology in the short term or any pathology not allowing participation in the study

Controls:

* Any clinical symptoms suggesting an acute infection
* Any life-threatening pathology in the short term or any pathology not allowing participation in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Performance at the 6 minute step-up test | Baseline, Month 6 and Month 12
  Number of ascent-descent cycles counted over 6 minutes

SECONDARY OUTCOMES:
Performance at the 6 minute walking test | Baseline and Month 12
  Distance covered during a 6-minute period of rapid walking on a flat and hard surface
Performances at the 6 minute stand up test | Baseline, Month 6
  Number of stand up - sit movements performed during a 6 minute period
Performances at the Y balance Test | Baseline
  Sum of distances reached in each direction (the best is chosen for each direction) divided by 3 x length of lower limb (standardization) and multiplied by 100
Grip strength | Baseline, Month 6 and Month 12
  Force in kg measured with a dynamometer, twice per limb
WHO Disability Assessment Schedule - 2.0 (WHODAS) score | Baseline and Month 12
  Score ranging between 0 and 100. Higher score indicates higher levels of difficulties for functioning
HIV Disability Questionnaire - short form (HDQ-SF) score | Day 0
  The higher the calculated score, the more significant the encountered difficulties
Short Physical Performance Battery (SPPB) score | Baseline and Month 12
  Score between 0 and 12, with 0 indicating the worst performance and 12 the highest degree of functionality
Scores of the Neuroscreen app tests | Baseline and Month 12
  Scores calculated by the application overall and for different cognitive domains: that higher scores indicated better performance.
Fasting blood glucose | Baseline and Month 12
  Measured on capillary blood
IDIR test | Baseline, Month 6 and Month 12
  Measure of urinary branched chain amino acid (BCCA) to detect insulin resistance
WHO-QoL | Baseline, Month 6 and Month 12
  Quality of life brief questionnaire (WHO). It includes 26 items measured on 5 point scales.
PHQ-9 | Baseline, Month 6 and Month 12
  Short questionnaire on depression. Score ranging from 0 to 27. Higher score indicates depressive symptoms
Satisfaction and acceptability of physical activity | Week 12, Month 6 and Month 12
  Questionnaire based on Sekhon's framework. Use 5-point Likert scales

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Debeaudrap, Principal Investigator — IRD; Patrick Coffie, Principal Investigator — PAC-CI
Locations (2):
- Côte d’Ivoire (2):
  - Centre Médical Spécialisé El Rapha, Abidjan
  - Formation semi urbaine (FSU) d'Abobo Avocatier, Abidjan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diadhiou N, Assoumou N, Tegbe J, Boa HE, Bao ML, Amador-Paz S, Vitiello D, Coffie P, Debeaudrap P. Effectiveness and Implementation of Adapted Physical Activity Delivery Strategies for Older Adults Living With HIV in Ivory Coast: Protocol for a Type 2 Hybrid Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 6;15:e84677. doi: 10.2196/84677. PMID 41494181